CLINICAL TRIAL: NCT05409729
Title: Evaluation of Ovarian Reserve in Women With Subclinical Hypothyrodism in Reproductive Age
Brief Title: Subclinical Hypothyrodism and Ovarian Reserve
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Ahmed Abed Eltawaab Abdo, Principal Investigator, Assiut University
Other Study IDs: AMH
Record Dates: First submitted 2022-06-04; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Fertility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: retrospective charts reviewing

SUMMARY:
This study aimed to evaluate the potential association of subclinical hypothyrodism and ovarian reserve in reproductive age in age groups more than 35 and age groups less than 35 using retrospective study included women with subclinical hypothyrodism and controls .Evaluation of potential association of antithyroid antibodies positivity on ovarian reserve

Primary outcome:

Measure the association of SCH with ovarian reserve markers (basal FSH ,LH/basal AFC /AMH)

DETAILED DESCRIPTION:
Thyroid dysfunction is one of the commonest disorders in women of reproductive age .there is association between subclinical hypothyrodism and infertility and ovarian reserve .It's known that subclinical hypothyrodism can be associated with reduced ovarian reserve in women more than 35 years old .Aclear association between subclinical hypothyrodism and ovarian reserve not established in reproductive age in women less than 35 .This retrospective study investigate serum thyroid hormone /Antithyroid hormone ,ovarian reserve markers (basal FSH,AMH,Antral follicle count on day 2-4/prolactin level .

ELIGIBILITY:
Inclusion Criteria:

* All reproductive age groups included women less than 35 and women more than 35

Exclusion Criteria:

* Previous ovarian surgery Women with long term thyroid hormone replacement Endometriosis History of radiotheraby

Ages: 13 Years to 45 Years | Sex: Female
Age Groups: Child, Adult
Study Population: patients with thyroid dysfunction who seeking fertility
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Measure the association of SCH with ovarian reserve markers (basal FSH ,LH/basal AFC /AMH) | 48 months
  This study aimed to evaluate the potential association of subclinical hypothyrodism and ovarian reserve in reproductive age in age groups more than 35 and age groups less than 35 using retrospective study included women with subclinical hypothyrodism and controls .Evaluation of potential association of antithyroid antibodies positivity on ovarian reserve

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Medical School, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rao M, Wang H, Zhao S, Liu J, Wen Y, Wu Z, Yang Z, Su C, Su Z, Wang K, Tang L. Subclinical Hypothyroidism Is Associated with Lower Ovarian Reserve in Women Aged 35 Years or Older. Thyroid. 2020 Jan;30(1):95-105. doi: 10.1089/thy.2019.0031. Epub 2019 Dec 20. PMID 31650898
- [Result] Korevaar TIM, Minguez-Alarcon L, Messerlian C, de Poortere RA, Williams PL, Broeren MA, Hauser R, Souter IC. Association of Thyroid Function and Autoimmunity with Ovarian Reserve in Women Seeking Infertility Care. Thyroid. 2018 Oct;28(10):1349-1358. doi: 10.1089/thy.2017.0582. Epub 2018 Aug 14. PMID 29943679